CLINICAL TRIAL: NCT06947434
Title: Effects of Laughter Yoga on Sexual Functioning, Anxiety, Depression, Fatigue, and Quality of Life in Patients With Multiple Sclerosis: A Quasi-Experimental Study
Brief Title: Laughter Yoga for Improving Sexual Function and Psychosocial Outcomes in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Cansu POLAT DÜNYA, PhD, Assistant Professor, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/352
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis; Sexual Dysfunction
Keywords: multiple sclerosis; sexual life; anxiety; depression; quality of life; laughter yoga
MeSH Terms: conditions — Multiple Sclerosis; Sexual Dysfunction, Physiological; Anxiety Disorders; Depression | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: This study utilizes a single-group pretest-posttest quasi-experimental design to evaluate the effects of a structured laughter yoga intervention on psychological symptoms (anxiety and depression), fatigue, sexual life, and quality of life in individuals with multiple sclerosis (MS). The model includes three data collection points: baseline (Week 0), five weeks after the pretest (Week 5, without intervention), and post-intervention (Week 11, after 10 laughter yoga sessions). This within-subject design allows for the comparison of participant outcomes over time, enabling the assessment of changes attributable to the intervention. No control group is included in this design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Participants in this single-arm study will undergo a structured laughter yoga intervention after a 5-week observation period without any intervention. The intervention consists of 10 sessions delivered over the subsequent 5 weeks (2 sessions per week). Each session lasts approximately 40 minutes and is conducted online via Zoom. Sessions include four core components: rhythmic clapping, deep breathing exercises (pranayama), playful activities, and guided laughter exercises.
  This design allows within-subject comparison of outcomes before and after the intervention. The goal is to assess the effects of laughter yoga on sexual functioning and psychological well-being in individuals with multiple sclerosis.
  Interventions: Other: Laughter Yoga

INTERVENTIONS:
Other: Laughter Yoga — Laughter yoga is a behavioral intervention that combines intentional laughter exercises with yogic breathing techniques. In this study, the intervention consisted of 10 sessions delivered over five weeks (two sessions per week), each lasting approximately 40 minutes. Sessions were conducted live via Zoom and included components such as rhythmic clapping, deep breathing (pranayama), playful movements, and guided laughter exercises. The aim was to promote relaxation, reduce stress, and enhance psychological well-being in individuals with multiple sclerosis.

SUMMARY:
The goal of this clinical trial is to evaluate whether laughter yoga can improve sexual functioning and reduce psychological symptoms in adults diagnosed with multiple sclerosis (MS). The main questions it aims to answer are:

Does laughter yoga improve sexual functioning in individuals with MS?

Does laughter yoga reduce anxiety, depression, and fatigue, and improve quality of life in this population?

Participants will:

Attend 10 online laughter yoga sessions over 5 weeks (2 sessions per week, 40 minutes each)

Complete online questionnaires before, during, and after the intervention to assess sexual functioning, anxiety, depression, fatigue, and quality of life

DETAILED DESCRIPTION:
This quasi-experimental study investigates the effectiveness of laughter yoga in improving sexual functioning and psychosocial outcomes in adults with multiple sclerosis (MS). Laughter yoga is a behavioral intervention combining voluntary laughter with yogic breathing techniques, aiming to enhance emotional well-being and reduce stress-related symptoms.

The study includes three assessment points: baseline (pretest), five weeks after the baseline (pre-intervention), and post-intervention. The intervention consists of 10 structured laughter yoga sessions conducted via Zoom over a 5-week period. Each session lasts approximately 40 minutes and includes rhythmic clapping, deep breathing exercises, playful activities, and simulated laughter practices guided by a certified laughter yoga facilitator.

Validated self-report instruments are used to assess sexual functioning, anxiety, depression, fatigue, and quality of life. The study specifically targets individuals with MS who report sexual problems and experience mild to moderate psychological symptoms.

The primary aim is to determine the effect of laughter yoga on sexual functioning (measured by MSISQ-19). Secondary outcomes include changes in anxiety, depression, fatigue, and health-related quality of life. This study seeks to explore laughter yoga as a feasible, non-pharmacological, and low-cost approach to improving multidimensional well-being in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosed with multiple sclerosis (MS)
* Literate and able to complete self-report questionnaires
* Expanded Disability Status Scale (EDSS) score < 4
* HADS-Anxiety score > 10
* HADS-Depression score > 7
* Reporting sexual problems based on MSISQ-19
* Having an active sexual life
* Access to internet and a device capable of video conferencing
* Willing to participate and able to attend all 10 laughter yoga sessions

Exclusion Criteria:

* MS relapse or acute exacerbation within the last 3 months
* Severe cognitive impairment or communication difficulties
* Current participation in any laughter therapy, yoga, or similar psychosocial intervention
* Diagnosis of a major psychiatric disorder (e.g., schizophrenia, bipolar disorder)
* Unwillingness or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Sexual Functioning (MSISQ-19 Total Score) | Baseline (Week 0), Pre-Intervention (Week 5), and Post-Intervention (Week 11)
  Sexual functioning will be assessed using the Multiple Sclerosis Intimacy and Sexuality Questionnaire-19 (MSISQ-19). This scale includes 19 items measuring primary, secondary, and tertiary sexual dysfunctions in individuals with MS. Scores range from 19 to 95, with higher scores indicating greater dysfunction. A reduction in score reflects improvement in sexual functioning.

SECONDARY OUTCOMES:
Change in Anxiety Level (HADS-A Score) | Baseline (Week 0), Pre-Intervention (Week 5), and Post-Intervention (Week 11)
  Anxiety levels will be measured using the Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A). Scores range from 0 to 21, with higher scores indicating greater anxiety. A decrease in the score reflects improvement.
Change in Fatigue Level (Fatigue Severity Scale Score) | Baseline (Week 0), Pre-Intervention (Week 5), and Post-Intervention (Week 11)
  Fatigue will be assessed using the Fatigue Severity Scale (FSS), consisting of 9 items rated on a scale from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater fatigue. A mean score ≥4 indicates clinically significant fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University School Of Nursing, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No